CLINICAL TRIAL: NCT07058441
Title: Clinical and Mechanistic Research on Autogenous Arteriovenous Fistula in Hemodialysis Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Ai Peng (Other)
Responsible Party: Sponsor-Investigator, Ai Peng, Director of the department of Nephrology, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: 25K118
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Arteriovenous Fistula Maturation Failure in End-stage Renal Disease
Keywords: Arteriovenous fistula maturation failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vascular tissues will be preserved for histopathological examination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single observational cohort of end-stage renal disease patients receiving initial autogenous arterio: This is an observational study with no investigational interventions. Standard clinical AVF surgical procedures will be performed per hospital protocols.

SUMMARY:
This study aims to investigate the long-term clinical outcomes and molecular mechanisms of autogenous arteriovenous fistula (AVF) maturation failure in uremic patients. The primary goal is to develop a precision prediction model integrating clinical, imaging, and biomarker data, while secondary objectives focus on identifying key molecular targets regulating AVF maturation.

DETAILED DESCRIPTION:
This observational study aims to investigate the long-term clinical outcomes and molecular mechanisms underlying autogenous arteriovenous fistula (AVF) maturation failure in uremic patients, with the primary goal of developing a precision prediction model integrating clinical, imaging, and biomarker data while also identifying key molecular targets regulating AVF maturation. Conducted as a single-center prospective study at Shanghai Tenth People's Hospital, the research will enroll 300 ESRD patients undergoing first-time AVF creation, collecting comprehensive multi-omics data including clinical parameters (demographics, comorbidities, laboratory tests), ultrasound imaging (vessel diameter, blood flow measurements), and molecular biomarkers (miRNAs, cytokines, vascular remodeling proteins). Using advanced machine learning techniques like Random Forest and XGBoost, the study will construct a predictive model for AVF maturation failure based on KDOQI criteria (blood flow <600 mL/min, diameter <6 mm, or depth >6 mm at 6 weeks), while parallel mechanistic investigations will employ WGCNA and Cox regression analyses to elucidate critical molecular pathways such as VEGF/TGF-β signaling and potential therapeutic targets including ALPL and Eph-B4. The study adheres to strict ethical guidelines (Helsinki Declaration, GCP standards) and includes rigorous statistical planning with a sample size calculated to ensure adequate power (300 patients yielding 110 expected events), employing AUC analysis for model discrimination and standard statistical tests for group comparisons. Expected outcomes include the development of a clinically applicable prediction tool (targeting software copyright), 2-3 high-impact SCI publications, and identification of novel therapeutic targets, with the entire project spanning from patient recruitment (2025.07-2026.07) through data analysis and manuscript preparation (2026.11-2027.01), ultimately aiming to significantly improve AVF management through its innovative combination of multi-omics integration and machine learning approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosed with chronic kidney disease stage 5 (ESRD) and scheduled for first-time autogenous AVF creation
3. No severe coagulation disorders or vascular malformations
4. Willing to provide written informed consent
5. Planned hemodialysis at the study center

Exclusion Criteria:

1. Previous AVF surgery on the ipsilateral limb
2. Ipsilateral central venous stenosis or significant venous outflow obstruction
3. Active malignancy (except localized non-melanoma skin cancer)
4. Active infection at the surgical site
5. Life expectancy <1 year
6. Pregnancy or lactation
7. Participation in other interventional trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll 300 adult ESRD patients undergoing initial autogenous arteriovenous fistula (AVF) creation at Shanghai Tenth People's Hospital. The population represents typical hemodialysis candidates with end-stage renal failure requiring vascular access. Participants will be recruited consecutively from nephrology and vascular surgery clinics, reflecting real-world clinical practice. The cohort will include patients with varied comorbidities (e.g., diabetes, hypertension) but exclude those with conditions that may confound AVF maturation assessment (prior access surgery, limited life expectancy). All patients will receive standard preoperative evaluation including vascular mapping ultrasound.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Arteriovenous fistula maturation failure rate | 6 weeks and 6 months post-surgery
  Failure to meet KDOQI criteria at 6 weeks post-operation (blood flow <600 mL/min, venous diameter <6 mm, OR subcutaneous depth >6 mm) AND inability to sustain hemodialysis (2 sessions/week)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology & Rheumatology, Shanghai Tenth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No